CLINICAL TRIAL: NCT05035732
Title: A Prospective Pilot Study for the Evaluation of 18F- Fluciclovine PET/MRI in Radio-recurrent Prostate Cancer (RRPC-PET/MRI Study)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0146; NCI-2021-09407 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer; Prostate Nodule
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-ACBC (Experimental)
  Interventions: Radiation: 18F-fluciclovine

INTERVENTIONS:
Radiation: 18F-fluciclovine — IV

SUMMARY:
To perform both PET scans and MRIs in the same setting using a simultaneous PET/MRI scanner.

DETAILED DESCRIPTION:
Primary Objective:

--To compare the diagnostic performance of 18F- Fluciclovine pelvic PET/MRI to that of pelvic mpMRI and to determine whether 18F- Fluciclovine pelvic PET/MRI is more accurate than a pelvic mpMRI in detecting pelvic RRPC in men with biochemical recurrence with histopathology as reference standard.

Secondary Objective:

--To study inter-reader reliability of 18F- Fluciclovine pelvic PET/MRI and pelvic mpMRI among the readers.

Exploratory Objective:

--To study correlation between SUVmax and ADCmean in the pelvic RRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients who are 18 years and older
2. Histologically or cytologically proven prostate carcinoma s/p definitive radiation
3. Patients suspected to have BCR based on phoenix criteria (prostate specific antigen value (PSA) of 2 ng/mL above the PSA nadir)
4. Ability to understand and willingness to sign informed consent

Exclusion Criteria:

1. Patients with any medical condition or circumstance that the investigator believes may compromise the data collected or lead to a failure to fulfil the study requirements.
2. Patients with contraindication to undergo MRI
3. Patients with prior allergy to MRI contrast agent.
4. Extreme Claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
To assess the diagnostic performance of 18F- Fluciclovine pelvic PET/MRI to that of pelvic mpMRI | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Devaki S Surasi, Principal Investigator — M.D. Anderson Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org